CLINICAL TRIAL: NCT02302027
Title: Feasibility Study of Normobaric Oxygen Delivered by a High Flow Concentrator in the Treatment of Chronic Headache With or Without Abuse of Painkillers
Brief Title: Feasibility Study of Normobaric Oxygen Delivered by a High Flow Concentrator in the Treatment of Chronic Headache
Acronym: O214
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association pour la Recherche au Centre d'Urgence des Céphalées (Other)
Responsible Party: Principal Investigator, Caroline ROOS, Medical Doctor, Association pour la Recherche au Centre d'Urgence des Céphalées
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARCUC
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Headache
Keywords: withdrawal therapy; oxygen therapy
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- platinium IRC9LXO2AWQ (Experimental): Normobaric oxygen therapy with high flow concentrator to treat headaches attacks, 30 minutes of oxygene inhalation with mask, 9l/minute, no frequency limitation
  Interventions: Device: platinium IRC9LXO2AWQ

INTERVENTIONS:
Device: platinium IRC9LXO2AWQ — high flow concentrator delivering normobaric oxygen after extraction, 9 liter per minute dimensions: 46 * 67 * 36 cm

SUMMARY:
Chronic headache is most often associated with drug abuse and medication overuse headache (MOH) is the main complication of migraine disease results in chronic daily headache. The first phase of treatment consists of drug withdrawal .

The second phase of treatment (called consolidation) is to maintain the balance: treating headaches and reducing / stopping the drug use.

The aim of this study is

1. verify the feasibility of a home withdrawal treatment with normobaric oxygen therapy (NOT) delivery by high flow concentrator
2. use normobaric oxygen therapy (NOT) as a therapeutic measure to treat headache through withdrawal period.

It is a feasibility pilot study in chronic headache with or without medication-overuse. All patients receive a care for outpatient withdrawal that involves sudden stop drug abuse and used to be called "traditional management". The subsequent attacks will be treated with NOT from a high-flow concentrator

Primary endpoint. Feasibility study of treatment with NOT evaluated by the percentage of patients who accepted NOT during the withdrawal phase then to treat attacks.

Secondary endpoints. Efficacy will be assessed by the percentage of patients having no chronic headaches two months after the start of withdrawal (less than 15 days of headache per month) and no longer in drug abuse (less than 10 days per month with drug intake).

Visits V1 (first visit) Inclusion V2 at one month V3 at 3 months V4 (last vist) at 6 months

Effective : 30 patients

ELIGIBILITY:
Inclusion Criteria:

* Migrainous according to the criteria of the International Headache Society
* Medication-overuse headaches according of the International Headache Society
* No prophylaxis treatment or same prophylaxis treatment from more than one month
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* One or more failed withdrawal treatment
* analgesic treatment for another reason than headache
* Contraindication of normobaric oxygen therapy
* Contraindication of ketoprofen (rescue therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
percentage of patients accepted the normobaric oxygen treatment during withdrawal and consolidation phases | 6th month

SECONDARY OUTCOMES:
number of headache days per month | 6th month
number of session of oxygen during the 6 months | 6th month
number of rescue medication taking on the 6 months | 6th month
Hospital Anxiety and Depression Scale | 1st month, 2d month and 3rd month
Headache Impact Test- 6 | 1st, 2d and 3rd month
Patient Global Impressions of Change Scale | 1st, 2d, 3rd, 4th, 5th and 6th month
Migraine Disability Assessment Questionnaire Scale | 3rd and 6th month

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Urgence des Céphalées, hôpital Lariboisière, Paris, France

REFERENCES:
- [Result] Kavuk I, Katsarava Z, Selekler M, Sayar K, Agelink MW, Limmroth V, Diener HC. Clinical features and therapy of medication overuse headache. Eur J Med Res. 2004 Dec 22;9(12):565-9. PMID 15689304
- [Result] Lanteri-Minet M, Valade D, Geraud G, Chautard MH, Lucas C. Migraine and probable migraine--results of FRAMIG 3, a French nationwide survey carried out according to the 2004 IHS classification. Cephalalgia. 2005 Dec;25(12):1146-58. doi: 10.1111/j.1468-2982.2005.00977.x. PMID 16305603
- [Result] Evers S, Marziniak M. Clinical features, pathophysiology, and treatment of medication-overuse headache. Lancet Neurol. 2010 Apr;9(4):391-401. doi: 10.1016/S1474-4422(10)70008-9. PMID 20298963